CLINICAL TRIAL: NCT01579669
Title: Partnering With Autistic Adults to Develop Tools to Improve Primary Healthcare
Brief Title: Partnering With Autistic Adults to Improve Healthcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Syracuse University (Other); Indiana University (Other); Autistic Self Advocacy Network (Unknown); Portland State University (Other)
Responsible Party: Principal Investigator, Christina M. Nicolaidis, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: R34MH092503 (NIH); R34MH092503 (NIH)
Record Dates: First submitted 2012-04-13; First posted 2012-04-18 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Primary Care Services; Patient-Provider Communication; Adults
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Use of Toolkit (Experimental): All participants will have access to the toolkit
  Interventions: Behavioral: Use of toolkit

INTERVENTIONS:
Behavioral: Use of toolkit — Patient participants will be given access to the toolkit and will create a customized report for their provider. Team will send report to providers and ask them to schedule appointment with patient to discuss.

SUMMARY:
The goal of this proposal is to develop and evaluate patient-centered care tools for autistic adults and their primary care providers (PCPs).

DETAILED DESCRIPTION:
The goal of this study is to develop and evaluate patient-centered care tools for autistic adults and their primary care providers (PCPs). One tool will allow autistic adults and/or their supporters to provide individualized information to PCPs about how being on the spectrum affects their healthcare and possible strategies to facilitate quality care. Another tool will capitalize on the power of patient narrative to educate PCPs about autism. These tools and other resources will be housed on an interactive website for autistic adults, supporters, and PCPs. The research team will evaluate the feasibility and acceptability of using the new web-based patient-centered care tools with autistic adults and their primary care providers. This study will provide data for a future trial testing the effectiveness of these tools in improving the health of autistic adults by increasing patient-centered care and patient activation.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of autism spectrum disorder (including autistic disorder, Asperger's disorder, Childhood Disintegrative Disorder, and pervasive developmental disorder NOS)
* Understands written or spoken English or has a support person available who understands written or spoken English
* Has a primary care provider

Exclusion Criteria:

* Is not a resident of the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Nicolaidis, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Nicolaidis C, Raymaker D, McDonald K, Kapp S, Weiner M, Ashkenazy E, Gerrity M, Kripke C, Platt L, Baggs A. The Development and Evaluation of an Online Healthcare Toolkit for Autistic Adults and their Primary Care Providers. J Gen Intern Med. 2016 Oct;31(10):1180-9. doi: 10.1007/s11606-016-3763-6. Epub 2016 Jun 6. PMID 27271730
- See also: AASPIRE toolkit study information — http://aaspire.org/?p=projects&c=hctoolkit/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited autistic adults via fliers, postings, and announcements targeted to autism and disability-related list-serves, organizations, and forums. We invited the autistic adult's primary care providers (PCPs) to participate if the patient gave permission for us to contact their provider and provided usable contact information.
Pre-assignment Details: The total number of participants enrolled includes everyone who consented to participate. Some participants clicked "yes" to the online consent, but did not participate in the initial survey. The number of participants noted as Started in the Participant Flow module includes only those that took the initial survey.
Groups:
- Autistic Adults: Adults on the autism spectrum
- Primary Care Providers: Participants' primary care providers
Period: Overall Study
Arm/Group | Autistic Adults | Primary Care Providers
Started | 170 | 41
Completed | 134 | 41
Not Completed | 36 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the autistic participants who completed the pre-intervention survey and the primary care providers who completed the PCP survey.
Groups:
- Primary Care Providers: Primary care providers taking care of autistic adults participating in this study
- Total: Total of all reporting groups
Arm/Group | Autistic Adults | Primary Care Providers | Total
Number analyzed (Participants) | 170 | 41 | 211
Age, Continuous [Mean (Full Range); unit: years] | 36.5 [18 to 68] | 36.3 [28 to 62] | 36.4 [18 to 68]
Sex/Gender, Customized [Number; unit: participants]
  Male | 75 | 15 | 90
  Female | 91 | 25 | 116
  Other | 4 | 0 | 4
  Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 1 | 12
  Not Hispanic or Latino | 158 | 36 | 194
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 152 | 29 | 181
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 170 | 41 | 211

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: Autistic participants completed an online survey about their satisfaction with the tool, including if they feel the tool is useful, how they think the tool will affect their healthcare, if and how they plan to use it with providers, and if they would recommend it to others.
Time Frame: 1 month after use of toolkit
Measure: Number; unit: percentage of participants
Arm/Group | Autistic Adults
Number analyzed (Participants) | 134
percentage of participants
  Percentage rating toolkit as useful | 95.08
  Percentage who felt toolkit was easy to use | 95.96
  Percentage who felt toolkit was important | 96.8
  Percentage who would recommend toolkit to friend | 92.11
  Percentage who would recommend toolkit to provider | 94.87

2. Secondary Outcome: Provider Satisfaction
Description: Providers participated in a brief survey to assess satisfaction with the toolkit. Items addressed overall satisfaction and if they would or would not use the tools with other patients.
Time Frame: 1-2 months after patient uses toolkit
Population: Participants' primary care providers. Primary care providers were included in the study to assess their impression of the toolkit, but all other outcomes (e.g. change in barriers, self-efficacy, or satisfaction with healthcare) only apply to the autistic participants, not their primary care providers.
Measure: Number; unit: percentage of PCPs
Arm/Group | Primary Care Providers
Number analyzed (Participants) | 41
percentage of PCPs
  Proportion rating AHAT as moderately or very usefu | 82.05
  Proportion who would recommend AHAT to patients | 86.49

3. Secondary Outcome: Patient Use of Toolkit Components
Description: We collected data on whether or not participants completed the Autism Healthcare Accommodations Tool (AHAT) survey and whether or not they allowed the research team to send a copy of the report to their primary care provider.
Time Frame: 1 month after use of toolkit
Measure: Number; unit: percentage of participants
Arm/Group | Autistic Adults
Number analyzed (Participants) | 170
percentage of participants
  Proportion completing AHAT | 96.00
  Proportion who requested AHAT be sent to provider | 57.74

4. Secondary Outcome: Change in Patient Satisfaction With Healthcare
Description: Patients completed an 8-item instrument assessing satisfaction with their primary healthcare experiences. The scale was previously adapted from the 2007 Health Information National Trends Survey (HINTS). In the pre-intervention survey autistic participants were asked to think about their last visit with their primary care provider. We did not assess patient-provider communication for those who were participating via a proxy as we did not feel that a proxy could adequately rate how satisfied the patient was with communication. Only autistic participants who said they had seen their PCP since using the healthcare toolkit were re-asked these items in the post-intervention survey. Responses used a 5-point Likert scale with anchors of "1 - Strongly Disagree" to "5 - Strongly Agree". We analyzed items by summing the responses into a composite score (range 8-40; higher scores indicate higher satisfaction). Cronbach's alpha = 0.92.
Time Frame: before and 1 month after use of toolkit
Population: Autistic adults who participated directly (not via a proxy) and who saw their provider in the 1 month between when they participated in the baseline assessment and they completed the post-intervention survey.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autistic Adults
Number analyzed (Participants) | 43
units on a scale
  Baseline Satisfaction | 30.91 (0.978)
  Post-intervention satisfaction | 32.63 (1.01)
Statistical Analysis 1: Comparison: Autistic Adults; Pre-post comparison; Test type: Superiority or Other; p = 0.0269, t-test, 2 sided

5. Secondary Outcome: Change in Patient's Perceived Barriers to Healthcare
Description: Autistic participants were presented with a list of 16 barriers to healthcare and asked which ones keep them from obtaining good care. We compared the total number of barriers endorsed by participants in the pre- and post-intervention surveys. The proxy version of the survey included a few modified items to differentiate between barriers faced by the autistic individuals and those faced by the supporter. Due to differences in the wording, we could not combine results from those who participated directly with those who participated by proxy. Only data from autistic adults who participated directly is shown.
Time Frame: Before and 1 month after use of toolkit
Population: Participants completing the pre and post-test themselves (not via a supporter).
Measure: Mean (Standard Error); unit: number of barriers
Arm/Group | Autistic Adults
Number analyzed (Participants) | 108
number of barriers
  Mean number of barriers at baseline | 4.07 (0.25)
  Mean number of barriers at follow-up | 2.82 (0.19)
Statistical Analysis 1: Comparison: Autistic Adults; Pre-post intervention comparison; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: Change in Patient Healthcare Self-Efficacy
Description: Autistic participants completed a 21-item healthcare self-efficacy scale before and 1 month after use of the toolkit. The scale was created de novo for this study, based on our prior qualitative work. Items addressed aspects related to healthcare navigation (e.g. "How confident are you that you can make an appointment with your healthcare provider when needed?"), successful interactions with providers, (e.g. "How confident are you that you can describe your symptoms or healthcare concerns to your provider?"), and self-management (e.g. "How confident are you that you can take medications the way you are supposed to take them?"). Response options used a 4-point Likert scale with anchors of "0 - Not at all confident" to "3 - Totally confident". We scored self-efficacy by adding responses from the 21 items, resulting in a possible range of 0 to 63, with higher scores corresponding to higher self-efficacy. Cronbach's alpha was 0.92.
Time Frame: Before and 1 month after use of toolkit
Population: Participants completing pre- and post-intervention survey themselves (not via a supporter), who had complete data on the self-efficacy scales on both surveys.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Autistic Adults
Number analyzed (Participants) | 98
units on a scale
  Baseline healthcare self-efficacy score | 37.92 (1.21)
  Follow-up healthcare self-efficacy score | 39.37 (1.19)
Statistical Analysis 1: Comparison: Autistic Adults; Pre-post intervention comparison; Test type: Superiority or Other; p = 0.016, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 month
Groups:
- Primary Care Providers: Primary care providers of autistic adults participating in the study.
Arm/Group | Autistic Adults | Primary Care Providers
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/41
Other Adverse Events (participants affected / at risk) | 0/170 | 0/41

LIMITATIONS AND CAVEATS:
This study was designed as a single-arm trial to assess feasibility and acceptability and to explore potential mechanisms of action. As such, there was no control group. PCPs are not a separate arm, but were included to assess acceptability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No